CLINICAL TRIAL: NCT05944432
Title: Real-Time Glucose Monitoring Using FreeStyle Libre 3 in Adults With Type 2 Diabetes On Basal Insulin Plus SGLT2 Inhibitor and/or GLP-1
Brief Title: CGM Use in Adults With Type 2 Diabetes on Basal Insulin
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADC-UK-PMS-22057
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FreeStyle Libre system (Active Comparator): FreeStyle Libre 3 continuous glucose monitoring system
  Interventions: Device: FreeStyle Libre 3 Continuous Glucose Monitoring System.
- Standard of care (control) (Other): Self monitoring of blood glucose
  Interventions: Device: Self monitoring of blood glucose

INTERVENTIONS:
Device: FreeStyle Libre 3 Continuous Glucose Monitoring System. — Subjects will be randomised to use the FreeStyle Libre 3 system
  Arms: FreeStyle Libre system
Device: Self monitoring of blood glucose — Subjects will be randomised to continue with their current glucose monitoring system
  Arms: Standard of care (control)

SUMMARY:
A prospective multi-centre, open-label, two arm, parallel design, superiority, pragmatic, randomised controlled trial, over an 8-month period. The purpose of this study is to determine whether continuous glucose monitoring using FreeStyle Libre 3 will improve HbA1c compared to SMBG over 16 weeks in adults with sub-optimally controlled (HbA1c 7.5-11%) Type 2 diabetes on basal therapy.

DETAILED DESCRIPTION:
The study will assess change in HbA1c as the primary endpoint. Other endpoints related to glycaemic control are included in the analyses. The study is split into two phases each of four months duration: participant-driven (phase 1) and HCP/therapy-driven (phase 2). Participants will be randomised to either FreeStyle Libre 3 or to continuation with their current SMBG device.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over.
* Type 2 diabetes diagnosis for ≥1 year prior to enrolment.
* Type 2 diabetes treated with a basal insulin injection regimen and SGLT2 inhibitor and/or GLP-1.
* Screening HbA1c ≥59 mmol/mol to ≤97 mmol/mol (≥7.5% and ≤11.0%, inclusive).

Exclusion Criteria:

* Participant is currently prescribed prandial or pre-mixed (biphasic) insulin at enrolment.
* Currently participating in another study that could affect glucose measurements or glucose management.
* A female participant who is pregnant.
* A breastfeeding female participant.
* Bariatric surgical procedure within the past 12 months or is planning/scheduled for bariatric surgery within the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  Difference between treatment groups in mean change from baseline in HbA1c.

SECONDARY OUTCOMES:
HbA1c | 32 weeks
  Difference between treatment groups in mean change from baseline in HbA1c
Time in range (TIR) | 32 weeks
  Time spent in glucose target range (TIR) 3.9 to 10.0 mmol/L (70 to 180 mg/dL).
Time above range (TAR) | 32 weeks
  Time spent above glucose target range (TAR) >10.0 mmol/L, 13.9 mmol/L and 16.7 mmol/L (>180 mg/dL, >250 mg/dL and >300 mg/dL).
Time below range(TBR) | 32 weeks
  Time spent below glucose target range (TBR) <3.9 mmol/L and <3.0 mmol/L (<70 mg/dL and <54 mg/dL).
Frequency of hypoglycaemia events | 32 weeks
  CGM detected hypoglycaemia events defined as ≥15 minutes duration with glucose <3.9 mmol/L (<70 mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Reid, Study Director — Abbott Diabetes Care Ltd
Locations (25):
- United Kingdom (25):
  - Tameside General Hospital, Ashton-under-Lyne
  - Royal United Hospital, Bath
  - Queen Elizabeth Hospital, Birmingham
  - Cambridge University Hospital (Addenbrookes), Cambridge
  - Darlington Memorial Hospital, Darlington
  - Royal Derby Hospital, Derby
  - Ninewells Hospital, Dundee
  - Princess Alexandra Hospital, Harlow
  - Northwick Park Hospital, Harrow
  - Hull Royal Infirmary, Hull
  - Ipswich Hospital, Ipswich
  - St James University Hospital, Leeds
  - Leicester General Hospital, Leicester
  - King's College Hospital, London
  - St Mary's Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Norfolk and Norwich University Hospital, Norwich
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - The Adam Practice, Poole
  - Queen Alexandra Hospital, Portsmouth
  - Northern General Hospital, Sheffield
  - Moorgreen Hospital, Southampton
  - Singleton Hospital, Swansea
  - Wishaw Hospital, Wishaw

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary study manuscript after deidentification (text, tables, figures and appendices) for the purposes of individual participant data meta-analysis.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 3 years (36 months) following article publication
Access Criteria: Researchers undertaking individual participant data meta-analysis who provide a methodologically sound proposal, approved by an independent review committee, and not overlapping with any planned secondary publications from the research team. Proposals should be directed to the corresponding author of the article who will discuss such requests with the study investigator team. To gain access, data requesters will need to sign a data access agreement. Data will be available for up to 3 years (36 months) following article publication.

REFERENCES:
- [Derived] Wilmot EG, Ajjan RA, Cheah YS, Choudhary P, Cranston I, Elliott RA, Evans M, Iqbal A, Kamaruddin S, Barnard-Kelly K, Lumb A, Min T, Moore P, Narendran P, Neupane S, Rayman G, Sathyapalan T, Thabit H, Yates T, Leelarathna L. Impact of real-time glucose monitoring using FreeStyle Libre 3 on glycaemia in type 2 diabetes managed with basal insulin plus SGLT2 inhibitor and/or GLP-1 agonist: the FreeDM2 randomised controlled trial protocol. BMJ Open. 2025 Apr 15;15(4):e090154. doi: 10.1136/bmjopen-2024-090154. PMID 40233956